CLINICAL TRIAL: NCT02073916
Title: Phase Ib Trial of Trastuzumab Emtansine In Combination With Lapatinib Plus Abraxane In Metastatic Her 2 Neu Over-Expressed Breast Cancer Patients
Brief Title: T-DM1 With Abraxane and Lapatinib for Metastatic HER2 Positive Breast Cancer
Acronym: STELA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jenny C. Chang, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jenny C. Chang, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009544; 0813-0139 (Other: HMRI IRB)
Record Dates: First submitted 2014-02-18; First posted 2014-02-27 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; HER2 positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Lapatinib; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T-DM1 + Lapatinib + Abraxane (Experimental): T-DM1 with Laptinib followed by Abraxane
  Interventions: Drug: T-DM1; Drug: Lapatinib; Drug: Abraxane

INTERVENTIONS:
Drug: T-DM1 — antibody-drug conjugate of trastuzumab and emtansine
  Other Names: Trastuzumab Emtansine; TE; Kadcyla
Drug: Lapatinib — Dual tyrosine kinase inhibitor (HER2 and EGFR)
  Other Names: Tykerb
Drug: Abraxane — albumin-bound paclitaxel. Chemotherapy - microtubule inhibitor
  Other Names: nab-paclitaxel

SUMMARY:
This open-label, single-center Phase Ib study will assess the safety and tolerability of combining trastuzumab emtansine (T-DM1) with Lapatinib and Abraxane in patients with metastatic HER2-positive breast cancer.

DETAILED DESCRIPTION:
This open-label, single-center Phase Ib study will assess the safety and tolerability of combining trastuzumab emtansine (T-DM1) with Lapatinib and Abraxane in patients with metastatic HER2-positive breast cancer. Patients will receive Abraxane on Day 1 of each 1-week cycle and T-DM1 on Day 1 of each 3-week cycle. Patients with take Lapatinib orally daily. Patients will receive the study treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented metastatic Her2 over-expressed breast cancer.
* Age ≥ 18 years Patients must have received at least two prior therapies for their malignant disease.
* Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)
* Adequate organ function (cardiac ejection fraction of ≥ 45%),
* CBC not less than .75 of institutional lower limit.
* Patients must have adequate liver function: AST and ALT < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis Bilirubin < 1.5 mg/dL
* Patients must have adequate renal function: creatinine <1.5 mg/dL is recommended; however, institutional norms are acceptable.
* Negative serum or urine β-hCG pregnancy test at screening for patients of childbearing potential
* Fertile patients must use effective contraception (barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed). Contraception method must be used during treatment and for three months after completing treatment Signed informed consent form (ICF)

Exclusion Criteria:

* Any medical or psychiatric condition that would prevent informed consent or limit survival to less than 4 weeks.
* Absolute QT interval of >460 msec in the presence of potassium >4.0mEq/L and Magnesium >1.8mg/dl.
* Patient with HIV and post- transplant associated lymphoproliferative disorders.
* Patient with concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of Trastuzumab Emtansine, Lapatinib or Abraxane.
* Pregnant or lactating women.
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab Emtansine, lapatinib, abraxane, or their components.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* Subjects with ulcerative colitis are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerable Dose | approximately 16 weeks
  Maximum tolerated dose (MTD) of Trastuzumab Emtansine in combination with Lapatinib plus Abraxane in metastatic Her2 over-expressed breast cancer.

SECONDARY OUTCOMES:
Dose Limiting Toxicities | From date of randomization through study follow up (approximately 16 weeks)
  Describe the dose-limiting toxicity (DLT) associated with Trastuzumab Emtansine in combination with Lapatinib plus Abraxane as assessed by CTCAE v4.0.
Measure toxicities associated with treatment combination | From date of randomization through study follow up (approximately 16 weeks)
  Describe and measure other toxicities associated with Trastuzumab Emtansine in combination with Lapatinib plus Abraxane as assessed by CTCAE v4.0.
Anti-tumor activity through imaging | approximately 16 weeks from randomization
  Document anti-tumor activity of Trastuzumab Emtansine in combination with Lapatinib plus Abraxane in metastatic Her2 over-expressed breast cancer as assessed by RECIST 1:1 criteria
Plasma pharmacokinetics and pharmacodynamic effect of treatment combination | Day 1 and 1,2,4,and 24hours
  Determine the plasma pharmacokinetics of Trastuzumab Emtansine in combination with Lapatinib plus Abraxane.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny C Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States